CLINICAL TRIAL: NCT00078065
Title: A Randomized Phase II Study of Xcellerated T CellsTM With or Without Prior Fludarabine Therapy in Patients With Multiple Myeloma
Brief Title: Xcellerated T CellsTM in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xcyte Therapies (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT005
Record Dates: First submitted 2004-02-18; First posted 2004-02-20 (Estimated); Last update posted 2005-11-11 (Estimated); Status verified 2005-03

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; fludarabine; Xcellerated T Cells
MeSH Terms: conditions — Multiple Myeloma

INTERVENTIONS:
Drug: Xcellerated T Cells

SUMMARY:
This trial is a phase II, randomized study of patients with multiple myeloma. All patients will receive Xcellerated T Cells, with or without prior fludarabine therapy.

15 patients in each study arm will be followed for 6 months.

DETAILED DESCRIPTION:
This randomized Phase II clinical study is designed to examine the safety and efficacy of Xcellerated T CellsTM, an activated, autologous T cell product, in subjects with multiple myeloma. Subjects must have failed at least one, but no more than three, prior cytotoxic therapies prior to study registration and may not have relapsed or progressed within one year following hematopoietic stem cell transplantation. Patients will be randomized to treatment with either Xcellerated T Cells alone, or lymphoablative therapy with fludarabine followed by Xcellerated T Cells. Thirty subjects will be treated, with 15 patients in each arm. Patients will be followed for six months following treatment.

ELIGIBILITY:
* Previous diagnosis of multiple myeloma (MM) based on standard criteria. Tests need not be performed within 30 days of registration.
* Failure of at least one, but no more than four, prior systemic therapies for MM prior to registration and may not have relapsed or progressed within 1 year following autologous hematopoietic stem cell transplantation. Repeat courses of the same therapeutic regimen separated in time by 6 or more months are considered separate therapies. Induction therapy followed by high dose chemotherapy and autologous hematopoietic stem cell transplantation counts as one therapy.
* Measurable serum and/or urine M-protein
* Disease progression or relapse, since most recent therapy for multiple myeloma
* Age > 18 years old and < 75 years old
* ECOG performance status of 0 or 1
* Females of child-bearing potential must have a negative serum bHCG test and be willing to use effective contraception (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the trial
* Negative test results for current/active infection with HIV-1, HIV-2, HTLV-1, HTLV-2, hepatitis B, and hepatitis C within 30 days of registration (Antibody, antigen, and nucleic acid tests acceptable, depending on institutional standards)
* Hemoglobin >= 10.0 g/dL. Transfusion with red blood cells or use of erythropoietin is permissible.
* White blood count (WBC) >= 3,000/mm3 and absolute neutrophil count (ANC) > 1000/mm3
* Platelet count > 75,000/mm3
* Corrected serum calcium < 11 mg/dL, and no evidence of symptomatic hypercalcemia. (Corrected serum calcium is calculated by adding 0.8 mg/dL to the measured serum calcium for every 1 g/dL that the serum albumin falls below 4.0 g/dL)
* Serum total bilirubin and alanine aminotransferase (ALT) < 2.0 times the upper limit of normal
* Serum creatinine < 2.5 mg/dL
* Serum human anti-mouse antibody (HAMA) titer undetectable or within the normal range, and no history of allergies to mice or murine (mouse) proteins
* The patient must be able to comprehend and have signed the informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-11; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Frohlich, MD, Study Chair — Xcyte Therapies
Locations (9):
- United States (9):
  - Oncotherapeutics, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Oregon Health Sciences University, Portland, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina